CLINICAL TRIAL: NCT05627102
Title: Structural and Functional Changes in Supraspinatus Tendinopathy Thtough Percutaneous Electrolysis and Neuromodulation Combined Therapy. A Single-blinded Randomized clínical Trial.
Acronym: EPTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Manuel Rodriguez Huguet, degree Physiotherapy, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPTE-NEUROMODULACIÓN
Record Dates: First submitted 2021-09-24; First posted 2022-11-25 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Supraspinatus Tendinitis
Keywords: tendinopathy; electrolysis; exercise; dry needling; physiotherapy
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: A specialist physician will be diagnosed the supraspinatus tendinopathy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Electrolysis and neuromodulation. (Experimental): The intervention for this group consisted of Therapeutic Percutaneous Electrolysis and neuromodulation. Patient received once week for four weeks associated with eccentric exercises device at home.
  Interventions: Other: Experimental Group
- Conventional group (Active Comparator): The multimodal physical therapy program includes 10 sessions of:
  ultrasound pulsatil therapy (US) for 10 minutes , transcutaneous electric nerve stimulation (TENS) for 20 minutes ans associated with eccentric exercises device at home.
  Interventions: Other: Conventional group

INTERVENTIONS:
Other: Experimental Group — Therapeutic Percutaneous Electrolysis an neuromodulation associated with eccentric exercises devices at home.
  Arms: Percutaneous Electrolysis and neuromodulation.
Other: Conventional group — Ultrasound pulsatil therapy (US), transcutaneous electric nerve stimulation (TENS) for 20 minutes and associated with eccentric exercises devices at home.
  Arms: Conventional group

SUMMARY:
The supraspinatus muscle tendinopathy show a big impact, however, there is a lack of awareness about the options of the physiotherapist treatment. It is necessary to do studies about effectiveness of therapeutic percutaneous electrolysis and neuromodulation. This technique enables treatment of the tendinopathies. To analyze the effectiveness of therapeutic percutaneou electrolysis and neuromodulation in the treatment of supraspinatus muscle tendinopathy. Single center randomized controlled trial, parallel treatment design. A specialist physician will be diagnosed the supraspinatus muscle tendinopathy. Participants will be randomly assigned to receive treatmen for 4 weeks: percutaneou electrolysis and neuromodulation associated with eccentric exercises or conventional treatment of Physiotherapy with the same eccentric exercises. Both interventions were performed under ultrasound guidance with a portable ultrasound (General Electric LogicE). Data will be collected by a blinded evaluator.

DETAILED DESCRIPTION:
Eccentric exercises of the supraspinatus muscle were performed in 3 sets of 10 repetitions. Participants were asked to perform the exercise program on an individual basis twice every day for 4 weeks. The eccentric program consisted of 3 exercises, focusing on the supraspinatus, infraspinatus, and scapular muscles. Participants were asked to do a normal abduction (concentric phase) and a slow return to the initial position (eccentric phase) included first the concentric phase, and the eccentric phase was slowly conducted. The exercise program was taught by a physiotherapist in the first session and monitored in the subsequent sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with supraspinatus tendinopathies that do not improve with conventional physiotherapy or pharmacological therapy protocols.
* Subjects who are in an active state of pain, who present painful symptoms in a sensitive and painful area of the tendon of insertion of the supraspinatus muscle in the humerus.

Exclusion Criteria:

* Individuals who have received surgery intervention in the same shoulder, or have suffered fractures or dislocations in the same shoulder.
* Individuals have received the proposed treatment in one month´s period previously.
* Individuals who suffering from cervical radiculopathies, fibromialgia síndrome, cardiac patients with pacemakers, cancer, infectious processes, or generalized lymphedema.
* Pregnant women can not receive this treatment intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The intensity of shoulder pain | Baseline
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).

SECONDARY OUTCOMES:
The intensity of shoulder pain | Four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
The intensity of shoulder pain | Twelve weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
The intensity of shoulder pain | twenty four weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of shoulder pain, and the worst and lowest level of pain experienced in the preceding week in the shoulder area. The minimal clinically important difference (MCID) for the NPRS in patients with shoulder pain was 1.1 points (Mintken, Glynn, and Cleland 2009).
Electromyographic activity | Baseline, four, twelve weeks and twenty four weeks.
  Electromyography (EMG) measures and records the electrical activity of a muscle.
Strength of The rotator cuff | Baseline, four, twelve weeks and twenty four weeks .
  The use of the hand dynamometer to measure the strength of shoulder movements
Questionnaire DASH. | Baseline, four, twelve weeks and twenty four weeks.
  Functionality in the arm.
Scale SPADI. | Baseline, four, twelve weeks and twenty four weeks.
  Functionality in the arm.
Assessment of structural changes in the tendon by ultrasound evaluation | Baseline, four, twelve weeks and twenty four weeks.
  Assessment of possible structural changes in the tendon by ultrasound evaluation of thickening, hypoechogenicity, and hypervascularity.

CONTACTS AND LOCATIONS:
Overall Officials: manuel manuel, Physiotherapy, Study Director — University of Cádiz
Locations (1):
- Manuel Rodríguez Huguet, Cadiz, Cádiz, Spain

REFERENCES:
- [Background] Cook JL, Purdam CR. Is tendon pathology a continuum? A pathology model to explain the clinical presentation of load-induced tendinopathy. Br J Sports Med. 2009 Jun;43(6):409-16. doi: 10.1136/bjsm.2008.051193. Epub 2008 Sep 23. PMID 18812414
- [Background] McCreesh K, Lewis J. Continuum model of tendon pathology - where are we now? Int J Exp Pathol. 2013 Aug;94(4):242-7. doi: 10.1111/iep.12029. PMID 23837792
- [Background] Khan KM, Cook JL, Maffulli N, Kannus P. Where is the pain coming from in tendinopathy? It may be biochemical, not only structural, in origin. Br J Sports Med. 2000 Apr;34(2):81-3. doi: 10.1136/bjsm.34.2.81. No abstract available. PMID 10786860
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Rodriguez-Huguet P, Ibanez-Vera AJ, Rodriguez-Almagro D, Martin-Valero R, Diaz-Fernandez A, Lomas-Vega R. Effectiveness of Percutaneous Electrolysis in Supraspinatus Tendinopathy: A Single-Blinded Randomized Controlled Trial. J Clin Med. 2020 Jun 12;9(6):1837. doi: 10.3390/jcm9061837. PMID 32545583
- [Background] Lewis JS. Rotator cuff tendinopathy. Br J Sports Med. 2009 Apr;43(4):236-41. doi: 10.1136/bjsm.2008.052175. Epub 2008 Sep 18. PMID 18801774
- [Background] Osborne JD, Gowda AL, Wiater B, Wiater JM. Rotator cuff rehabilitation: current theories and practice. Phys Sportsmed. 2016;44(1):85-92. doi: 10.1080/00913847.2016.1108883. Epub 2015 Nov 7. PMID 26548634
- [Background] Garcia Bermejo P, De La Cruz Torres B, Naranjo Orellana J, Albornoz Cabello M. Autonomic Responses to Ultrasound-Guided Percutaneous Needle Electrolysis: Effect of Needle Puncture or Electrical Current? J Altern Complement Med. 2018 Jan;24(1):69-75. doi: 10.1089/acm.2016.0339. Epub 2017 Jan 30. PMID 28135129
- [Background] Rodriguez-Huguet M, Gongora-Rodriguez J, Lomas-Vega R, Martin-Valero R, Diaz-Fernandez A, Obrero-Gaitan E, Ibanez-Vera AJ, Rodriguez-Almagro D. Percutaneous Electrolysis in the Treatment of Lateral Epicondylalgia: A Single-Blind Randomized Controlled Trial. J Clin Med. 2020 Jul 1;9(7):2068. doi: 10.3390/jcm9072068. PMID 32630241
- [Background] Littlewood C, Ashton J, Chance-Larsen K, May S, Sturrock B. Exercise for rotator cuff tendinopathy: a systematic review. Physiotherapy. 2012 Jun;98(2):101-9. doi: 10.1016/j.physio.2011.08.002. Epub 2011 Oct 5. PMID 22507359
- [Background] Dejaco B, Habets B, van Loon C, van Grinsven S, van Cingel R. Eccentric versus conventional exercise therapy in patients with rotator cuff tendinopathy: a randomized, single blinded, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2017 Jul;25(7):2051-2059. doi: 10.1007/s00167-016-4223-x. Epub 2016 Jun 28. PMID 27351548
- [Background] Heron SR, Woby SR, Thompson DP. Comparison of three types of exercise in the treatment of rotator cuff tendinopathy/shoulder impingement syndrome: A randomized controlled trial. Physiotherapy. 2017 Jun;103(2):167-173. doi: 10.1016/j.physio.2016.09.001. Epub 2016 Sep 21. PMID 27884499
- [Background] Kinsella R, Cowan SM, Watson L, Pizzari T. A comparison of isometric, isotonic concentric and isotonic eccentric exercises in the physiotherapy management of subacromial pain syndrome/rotator cuff tendinopathy: study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2017 Nov 14;3:45. doi: 10.1186/s40814-017-0190-3. eCollection 2017. PMID 29163981
- [Background] Lin ML, Chiu HW, Shih ZM, Lee PY, Li PZ, Guo CH, Luo YJ, Lin SC, Lin KY, Hsu YM, Pang A, Pang W. Two Transcutaneous Stimulation Techniques in Shoulder Pain: Transcutaneous Pulsed Radiofrequency (TPRF) versus Transcutaneous Electrical Nerve Stimulation (TENS): A Comparative Pilot Study. Pain Res Manag. 2019 Feb 4;2019:2823401. doi: 10.1155/2019/2823401. eCollection 2019. PMID 30863472
- [Background] Gunay Ucurum S, Kaya DO, Kayali Y, Askin A, Tekindal MA. Comparison of different electrotherapy methods and exercise therapy in shoulder impingement syndrome: A prospective randomized controlled trial. Acta Orthop Traumatol Turc. 2018 Jul;52(4):249-255. doi: 10.1016/j.aott.2018.03.005. Epub 2018 Apr 25. PMID 29703659
- [Background] Desmeules F, Boudreault J, Roy JS, Dionne C, Fremont P, MacDermid JC. The efficacy of therapeutic ultrasound for rotator cuff tendinopathy: A systematic review and meta-analysis. Phys Ther Sport. 2015 Aug;16(3):276-84. doi: 10.1016/j.ptsp.2014.09.004. Epub 2014 Sep 23. PMID 25824429
- [Background] Balci TO, Turk AC, Sahin F, Kotevoglu N, Kuran B. Efficacy of therapeutic ultrasound in treatment of adhesive capsulitis: A prospective double blind placebo-controlled randomized trial. J Back Musculoskelet Rehabil. 2018;31(5):955-961. doi: 10.3233/BMR-150482. PMID 30040706